CLINICAL TRIAL: NCT05840744
Title: Evaluation of Risk Factors, Clinical Pattern and Outcome of Thrombosis in Children
Brief Title: Evaluation of Risk Factors and Outcome of Thrombosis in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Haidy Abdelazim Youssif, Resident of pediatric and neonatology department, Sohag University Hospitals, Sohag University
Other Study IDs: Soh-Med-23-04-17MS
Record Dates: First submitted 2023-04-12; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Thrombosis in Children
MeSH Terms: interventions — Blood Cell Count; Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: complete blood count — Investigations done for identifying the risk factor which lead to thrombosis.
  Other Names: blood culture; CRP; Anti thrombin 3 if thrombophilia suspected

SUMMARY:
Pediatric thrombosis is multifactorial, and usually risk factors either congenital or acquired are present.

Patient may has one risk factor or more such as sepsis, cancers, congenital heart disease, post surgery , central venous catheter insertion, nephrotic syndrome, systemic lupus erythromatosis and inflammatory bowel disease.

If there's no obvious risk factor for thrombosis, hereditary thrombophilia is suspected which results when an inherited factor, such as antithrombin , protein C or protein S deficiency.

DETAILED DESCRIPTION:
Thrombosis is the formation of a blood clot (partial or complete blockage) within blood vessels, whether venous or arterial, limiting the natural flow of blood and resulting in clinical sequela.

Incidence of childhood thrombosis is 0.07-0.14/10,000 in the general population. This incidence has been reported to be 5.3/10,000 in children presenting to hospital, 0.51/10,000 in all newborns and 0.24/10,000 in children in neonatal intensive care units . Pediatric thrombosis is multifactorial, and usually risk factors either congenital or acquired are present. . Patient may has one risk factor or more such as sepsis, cancers, congenital heart disease, post surgery , central venous catheter insertion, nephrotic syndrome, systemic lupus erythromatosis and inflammatory bowel disease. If there's no obvious risk factor for thrombosis, hereditary thrombophilia is suspected which results when an inherited factor, such as antithrombin , protein C or protein S deficiency.

There are three changes described by Virchow in 1856 are involved in the formation of thrombosis:

1. Changes in blood flow (rheology, stasis)
2. Changes in the vascular wall
3. Changes in the blood levels of coagulation factors The diagnosis of thrombosis is made more frequently and more easily in children due to noninvasive diagnos-tic methods [Doppler and ultrasonography (US), echo-cardiography, computed tomography (CT) and magnet-ic resonance imaging (MRI)]. The morbidity and mortality rates are high, although it occurs more rarely compared with adult thrombosis and does not develop in the absence of a triggering factor; the rate of mortality related with direct venous thromboembolism is 2.2%, the frequency of post-thrombotic syndrome is 12.4%, and the recurrence rate for thrombosis is 8.1%.

ELIGIBILITY:
Inclusion Criteria:• All children age from one day to 18 yrs presented with any vascular thrombosis decomented by clinical picture and venous doppler study or radiological study.

-

Exclusion Criteria:

* • Persons above 18 years old.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: • All children age from one day to 18 yrs presented with any vascular thrombosis decomented by clinical picture and venous doppler study or radiological study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-04-13 (Estimated); Study Completion 2024-04-13 (Estimated)

PRIMARY OUTCOMES:
occurance of in-hospital mortality | 12 months
  detection the mortality occurance in patients with thrombosis within admission in hospital
Occurance of neurological deficit | 12 months
  occurance of neurological deficit at the end of hospital admission and before discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt